CLINICAL TRIAL: NCT01590745
Title: A Randomised Controlled Double Blind Trial Of Therapeutic Ultrasound in Carpal Tunnel Syndrome (CTS)
Brief Title: Ultrasound Therapy for Carpal Tunnel Syndrome (CTS)
Acronym: CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Kamalakannan Jothi, Highly Specialised Clinical Physiologist - Neurophysiology, East Kent Hospitals University NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011/NEURO/04/EKHT
Record Dates: First submitted 2012-04-26; First posted 2012-05-03 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Ultrasound therapy; Nerve Conduction studies; Boston and Levine Questionnaire; Neutral Angle Wrist Splint; Canterbury CTS scale
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Ultrasound regimen (Placebo Comparator): A switch in the transducer circuit allows mock ionisation as a result no ultrasound emitted.
  Interventions: Device: EMS Therasonic 460 Primo Ultrasound therapy
- Real Ultrasound therapy (Active Comparator): Pulsed mode ultrasound therapy
  Interventions: Device: EMS Therasonic 460 Primo Ultrasound therapy

INTERVENTIONS:
Device: EMS Therasonic 460 Primo Ultrasound therapy — 1MHz / 1.0W/cm square probe for 15 minutes per session for 20 sessions.
  Other Names: Ultrasound treatment

SUMMARY:
Carpal Tunnel Syndrome (CTS) is a recognisable pattern of symptoms and signs, which are caused by compression of the median (middle) nerve as it passes through the carpal tunnel at the wrist.

This condition affects individuals by causing pain, numbness, tingling sensations and sometimes weakness in the fingers and may extend to shoulder and neck areas. The cause for most cases is unknown (idiopathic) though some common conditions are associated with an increased incidence, including obesity, pregnancy, hypothyroidism, arthritis, diabetes, and trauma.

Diagnosis is primarily clinical and the condition is easily recognised from the characteristic symptoms in straightforward cases but diagnostic support is provided by investigations such as nerve conduction studies and ultrasound imaging.

Treatment may include splinting, local steroid injection at wrist, activity modification,physical or occupational therapy (controversial), medications, and surgery. Treatment with local therapeutic ultrasound has been suggested to be effective but existing trials are inconclusive.

Wrist splinting is only partially effective with a success rate of 34%, Steroid injection is followed by frequent relapses and there remains uncertainty about the safety of serial injections. Surgery is effective but has a small but significant incidence of permanent complications. Any demonstrably effective and safe addition to the therapeutic options would be a significant advance in treatment. Therapeutic ultrasound at present appears a promising option, having a very good safety record but so far uncertain evidence of efficacy.

In our trial patients, with mild carpal tunnel syndrome, confirmed by nerve conduction studies, will all be given wrist splints so that no patients will be left untreated. They will be randomly allocated to either therapeutic or sham ultrasound therapy (20 sessions over 7 weeks) and followed up for 1year. The patients, operators of the ultrasound equipment and assessors will all be blind to treatment allocation.

The effect of treatment on symptoms will be assessed using a validated questionnaire and nerve conduction studies will be repeated at completion of the ultrasound treatment, 6 and 12 months.

This study is designed to find out to whether therapeutic ultrasound is an effective treatment for carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the commonest peripheral nerve disorder in the UK. Average annual incidences (per 100 000) were 139.4 for women and 67.2 for men in East Kent, UK.

It has significant economic impact, on average having the largest recuperation period of all injuries / illness that require days away from work. It causes tingling, numbness or pain in the distribution of the median nerve (the thumb, index, and middle fingers, and half the ring finger) that is often worse at night and causes wakening. The pathology of idiopathic CTS is a non-inflammatory fibrosis of the subsynovial connective tissue surrounding the flexor tendons but the causes are not fully understood.

Many treatments have been proposed but reviews performed by the Cochrane collaboration have found firm evidence in support of only:

1. Surgical decompression of the carpal tunnel.
2. Steroid therapy (local injection or systemic administration).
3. Neutral angle wrist splinting.

None of the available evidence based treatments for CTS are entirely satisfactory. Splinting is only partially effective with a success rate of 34%, Steroid injection is followed by frequent relapses and there remains uncertainty about the safety of serial injections. Surgery results in a small but significant incidence of permanent morbidity from complications.

Any demonstrably effective and safe addition to the therapeutic options would be a significant advance. Of the many candidate treatments, therapeutic ultrasound at present appears the most promising and is therefore the subject of this proposal Therapeutic ultrasound has a very good safety record and is essentially non-invasive.

In this trial, patients with mild carpal tunnel syndrome, confirmed by nerve conduction studies, will all be given wrist splints. They will be randomly allocated to either real or sham ultrasound therapy (20 sessions over 7 weeks) and followed up for 1 year. The effect of treatment on symptoms will be assessed using a validated questionnaire and nerve conduction studies will be repeated at completion of the ultrasound treatment at 7th week and further after 6 and 12 months time.

This will be a randomised, double blind, single-centre, clinical trial conducted by East Kent Hospitals University Foundation Trusts (Kent and Canterbury Hospital), with follow-up for 1 year from completion of treatment. Following randomisation, patients will be required to attend the clinic for 20 sessions over a 7 weeks period (5x weekly for 2 weeks then 2x weekly for 5 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged between 18 and 90 years with mild carpal tunnel syndrome (Canterbury NCS grades 1-3).
* No Previous treatment history other than splinting and use of over the counter NSAIDs.

Exclusion Criteria:

* Subjects diagnosed with peripheral neuropathy, secondary entrapment neuropathies diabetes mellitus, rheumatoid disease, acute trauma.
* Previous carpal tunnel surgery.
* Pregnancy or lactating.
* Patients with known HIV infection.
* Other serious medical or psychiatric illness currently ongoing, or experienced within the past three months, that in the opinion of the investigator would compromise the study.
* Patients unable to comply with the protocol requirements, including severe alcohol and drug use.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Changes in Boston/Levine subjective Symptom score | Baseline, 7th week, 6 months and end of 12months
  Improvement in the Boston/Levine subjective Symptom score at completion of Ultrasound treatment(real or sham), a decrease of at least 1.04 points being considered a clinically significant change.

SECONDARY OUTCOMES:
Functional status score | 7th week, 6 months and end of 12 months
  Improvement in functional status score, participants overall opinion of outcome, duration of Ultrasound therapy effect and relapses will be assessed for one year.
Nerve Conduction Studies | Baseline,7th week, 6 months and end of 12 months
  Changes in Nerve Conduction Studies grading.
Ultrasound Imaging of Wrist(s) | Baseline, 7th week, 6 and 12 months
  Measurements of Cross section Area (CSA)of the median nerve at the wrist(s).

CONTACTS AND LOCATIONS:
Overall Officials: Kamalakannan Jothi, Principal Investigator — East Kent Hospitals University NHS Foundation Trust; Jeremy Bland, Study Chair — East Kent Hospitals University NHS Foundation Trust
Locations (1):
- East Kent Hospitals University NHS Foundation Trusts, Canterbury, Kent, United Kingdom

REFERENCES:
- [Background] Oztas O, Turan B, Bora I, Karakaya MK. Ultrasound therapy effect in carpal tunnel syndrome. Arch Phys Med Rehabil. 1998 Dec;79(12):1540-4. doi: 10.1016/s0003-9993(98)90416-6. PMID 9862296
- [Background] Ebenbichler GR, Resch KL, Nicolakis P, Wiesinger GF, Uhl F, Ghanem AH, Fialka V. Ultrasound treatment for treating the carpal tunnel syndrome: randomised "sham" controlled trial. BMJ. 1998 Mar 7;316(7133):731-5. doi: 10.1136/bmj.316.7133.731. PMID 9529407
- [Background] O'Connor D, Marshall S, Massy-Westropp N. Non-surgical treatment (other than steroid injection) for carpal tunnel syndrome. Cochrane Database Syst Rev. 2003;2003(1):CD003219. doi: 10.1002/14651858.CD003219. PMID 12535461
- [Background] Bland JD. A neurophysiological grading scale for carpal tunnel syndrome. Muscle Nerve. 2000 Aug;23(8):1280-3. doi: 10.1002/1097-4598(200008)23:83.0.co;2-y. PMID 10918269
- [Background] Bland JD, Rudolfer SM. Clinical surveillance of carpal tunnel syndrome in two areas of the United Kingdom, 1991-2001. J Neurol Neurosurg Psychiatry. 2003 Dec;74(12):1674-9. doi: 10.1136/jnnp.74.12.1674. PMID 14638888
- [Background] Bland JD. Do nerve conduction studies predict the outcome of carpal tunnel decompression? Muscle Nerve. 2001 Jul;24(7):935-40. doi: 10.1002/mus.1091. PMID 11410921
- [Background] Banta CA. A prospective, nonrandomized study of iontophoresis, wrist splinting, and antiinflammatory medication in the treatment of early-mild carpal tunnel syndrome. J Occup Med. 1994 Feb;36(2):166-8. doi: 10.1097/00043764-199402000-00012. PMID 8176515
- [Background] Foley JL, Little JW, Vaezy S. Effects of high-intensity focused ultrasound on nerve conduction. Muscle Nerve. 2008 Feb;37(2):241-50. doi: 10.1002/mus.20932. PMID 18041054
- See also: Click here for more information about carpal tunnel syndrome and canterbury patients can keep in touch with specialist through this web page. — http://www.carpal-tunnel.net/